CLINICAL TRIAL: NCT04186130
Title: Fecal Microbium Change in Pediatric Patients With Spina Bifida: Prospective Case-control Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0904
Record Dates: First submitted 2019-10-16; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Spina Bifida
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SB: Children over 3 years old and under 12 years old who have been diagnosed with spinal bifida with spinal MRI. They should not have known inflammatory bowel disease or cloacal anomaly
- Control: Children over 3 years old and under 12 years without known inflammatory bowel disease or cloacal anomaly

SUMMARY:
Purpose: In order to verify the hypothesis that the composition of intestinal microbiota in children with spina bifida is different from that of normal control, prospective comparative analysis would be performed.

Background of the study:

Spina bifida is a congenital neurological disorder, causing neurogenic bowel. It has been known that the intestinal microbiota in spinal cord injury patient was different than that of control. Changes in intestinal motility, mucous secretion, immune surveillance, and epithelial barrier permeability are possible causes of this change. As spina bifida is also related with neurogenic bowel, the investigators hypothesized that the intestinal microbiota in spina bifida is different from that of normal control.

Patients total 30 patients and 10 controls Inclusion for patients

Patients who meet following conditions:

1) Children over 3 years old and under 12 years old who have been diagnosed with spinal bifida with spinal MRI Exclusion for patients and controls

1) Children with known inflammatory bowel disease or cloacal anomaly

Statistical analysis Statistical processing for fecal samples is aimed at alpha or beta diversity using bioinformatics, and the Kruskal-Wallis test is used to compare similarities or differences between each fecal sample. Prior to statistical analysis, the relative abundance of the detected microorganisms is analyzed first, and microorganisms having a distribution less than 0.1% are excluded from the analysis, and the remaining microorganisms are analyzed in the 'genus' step.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children aged 3-12 years, diagnosed with spina bifida in spinal MRI.

Exclusion Criteria:

* 1. The patient has an inflammatory intestinal disease known in the colon or has a cloacal anomaly.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
the alpha or beta diversity of intestinal microbiota composition in children with spina bifida is different from that of normal control | 1 year
  Feces are collected about 1-2 grams and stored at -80'c refrigerator. After analysis, using biometrics, statistical processing for fecal samples is aimed at alpha or beta diversity. The Kruskal-Wallis test is used to compare similarities or differences between each fecal sample. Prior to statistical analysis, the relative abundance of the detected microorganisms is analyzed first, and microorganisms having a distribution less than 0.1% are excluded from the analysis, and the remaining microorganisms are analyzed in the 'genus' step.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No